CLINICAL TRIAL: NCT07291596
Title: The Effect of Foot-Ankle Exercises on Pain, Sleep Quality and Depression in Individuals With Diabetic Peripheral Neuropathy
Brief Title: Exercise Effects on Pain, Sleep and Depression in Diabetic Peripheral Neuropathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025000073
Record Dates: First submitted 2025-11-25; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: diabetes; neuropathy; Exercise; Pain; Sleep Quality; Depression
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity; Pain; Sleep Initiation and Maintenance Disorders; Depression

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled experimental type.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): This group will receive foot-ankle exercises 3 days a week, 2 times a day for 8 weeks.
  Interventions: Behavioral: Ankle-Foot Exercise Program
- Control Group (No Intervention): No intervention will be performed in this group. Individuals will receive their routine care.

INTERVENTIONS:
Behavioral: Ankle-Foot Exercise Program — A structured ankle-foot exercise program consisting of walking warm-up, ankle dorsiflexion and plantarflexion, hamstring stretching, toe and heel raises, towel-grasp toe exercise, and rolling massage with a spiky roller. Exercises will be performed 3 times per week, twice per day, for 8 weeks.
  Arms: Exercise Group

SUMMARY:
It is known that the pain experienced by individuals with diabetic neuropathy negatively impacts sleep and quality of life, leading to numerous psychosocial problems such as anxiety and depression. Studies in the literature indicate that exercise, a non-pharmacological method, improves pain and sleep quality in individuals with diabetic neuropathy. However, no studies have been found evaluating the effects of foot-ankle exercises on pain, sleep quality, and depression in individuals with diabetic neuropathy.

This research aims to examine the effects of foot-ankle exercises on pain, sleep quality, and depression in individuals with diabetic peripheral neuropathy.

This randomized controlled experimental study will be conducted with 70 individuals with diabetes diagnosed with diabetic neuropathy, registered in the patient information systems of two public hospitals. The foot-ankle exercises will be performed by the patients in their homes, twice a day, three days a week, for eight weeks. The research data are as follows: The Introductory Information Form will be collected using the S-Lanns (Self-Leeds Assessment of Neuropathic Symptoms and Sign) Pain Scale, VAS-Visual Analog Scale, Pittsburgh Sleep Quality Index (PSQI), and Beck Depression Inventory (BDI).

This study is important because it will determine the effects of foot and ankle exercises on pain, sleep disturbances, and depression, which are common problems experienced by individuals with diabetic neuropathy.

DETAILED DESCRIPTION:
Diabetic neuropathy affects approximately 50% of individuals with diabetes throughout their lives. Diabetic neuropathy accounts for approximately 30-50% of all neuropathy diagnoses. Diabetic neuropathy is classified according to the affected area. Peripheral involvement describes involvement of the lower or upper extremities. Peripheral involvement is more common than involvement of other areas, with a prevalence of 16-87% in individuals with diabetes. Individuals with diabetic peripheral neuropathy typically present to the hospital with numbness, tingling, pain, and loss of sensation in the extremities.

The symptoms experienced in diabetic neuropathy negatively impact individuals' quality of life, and pain is one of the most common symptoms. Diabetic neuropathic pain can be spontaneous, constant, or intermittent, and can be described as burning, stinging, tingling, numbness, or coldness, and can be localized to one or more areas. Neuropathic pain generally worsens at night and is more common in the feet.

Management of diabetic neuropathy includes the use of pharmacological agents, glycemic control, lifestyle changes, risk factor management, assessment of foot ulcer risk, foot care, and non-pharmacological interventions.

Non-pharmacological treatment methods have been shown to be effective in reducing pain and improving quality of life. These include transcutaneous electrical nerve stimulation, spinal cord stimulation, transcranial magnetic stimulation, reflexology, aromatherapy massage, spa treatments, and exercise.

Exercises are also included among the treatment methods.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Diagnosed with diabetic peripheral neuropathy for at least 6 months S-LANSS pain score ≥ 12
* Able to perform the exercise program
* Voluntary participation and informed consent

Exclusion Criteria:

* Pregnancy
* Severe cardiovascular or musculoskeletal disease
* Cognitive impairment preventing participation
* Receiving physiotherapy or another structured exercise program during the study
* Any other condition deemed inappropriate by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-12-22 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale for Pain | Baseline and 8 weeks.
  Pain severity will be assessed using the Visual Analog Scale for Pain, a 10-cm line on which participants rate their pain intensity from 0 to 10, where 0 indicates "no pain" and 10 indicates "worst imaginable pain." Higher scores represent more severe pain.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | Baseline and 8 weeks.
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI), which includes 19 items, of which 18 contribute to scoring across seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Each item is rated from 0 to 3, and component scores are summed to yield a global score ranging from 0 to 21. Higher scores indicate poorer sleep quality.
Self-report Leeds Assessment of Neuropathic Symptoms and Signs Pain Scale | Baseline and 8 weeks.
  Neuropathic pain will be evaluated using the Self-report Leeds Assessment of Neuropathic Symptoms and Signs (S-LANSS) Pain Scale, which includes 7 items. The first five items assess neuropathic pain symptoms, and the last two items assess the presence of allodynia and reduced pain sensation. Items are scored as "yes/no," producing a total score between 0 and 24. Scores ≥12 support neuropathic pain, while scores <12 suggest nociceptive pain. Higher scores indicate greater neuropathic pain severity.
Beck Depression Inventory | Baseline and 8 weeks.
  Depression severity will be measured using the Beck Depression Inventory (BDI), a 21-item self-report instrument that assesses cognitive, affective, and somatic symptoms. Each item is scored from 0 to 3, producing a total score that ranges from 0 to 63. Higher scores indicate more severe depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Çayır Yılmaz, PhD, Principal Investigator — Amasya University
Locations (1):
- Amasya University Sabuncuoğlu Şerefeddin Education and Research Hospital-Suluova State Hospital, Amasya, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be shared. Only the full thesis text (PDF) will be available through the YÖK National Thesis Center after completion.